CLINICAL TRIAL: NCT06377111
Title: Phase 1 Trial of PANtoTHEnic Acid in Patient With Metastatic or Unresectable Melanoma ON ImmunOtherapy (PANTHEON-IO)
Brief Title: A Study to Test the Benefit of Vitamin B5 in Patients With Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANTHEON-IO
Record Dates: First submitted 2024-04-05; First posted 2024-04-22 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Melanoma (Skin)
Keywords: Vitamin B5; Unresectable melanoma; Metastatic melanoma; Pantothenic acid; Combined immune checkpoint inhibitors; ICI; Nivolumab; Ipilimumab; Anti-PD-1 antibody; Anti-CLTA-4 antibody; Skin cancer; Melanoma; Calcium pantothenate
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Pantothenic Acid; Nivolumab; spartalizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-PAN in combination with ICI (Experimental): C-PAN will be taken orally once daily in the morning prior to eating. The daily oral dose of C-PAN is 2000 mg (4 capsules of 500 mg each). Subjects will receive C-PAN exclusively for a run-in period of 3 to 7 days, and then a maintenance dose as long as the patient continues to receive SOC Nivolumab and Ipilimumab. Treatment will continue until unacceptable toxicity, progression of disease (PD), start of new anticancer therapy, or for a maximum of 1 year, whichever occurs earlier, and in the absence of criteria to discontinue C-PAN.
  Interventions: Dietary Supplement: C-PAN; Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Dietary Supplement: C-PAN — C-PAN is an essential nutrient as it is required for the synthesis of CoA, a key cofactor in the tricarboxylic acid cycle and fatty acid metabolism, as well as for the synthesis of acyl carrier protein. Pantothenate appears to be safe in humans with studies describing the administration of doses up to 10 grams per day over prolonged periods of time; hence, no upper limit for tolerability has been established. In this study, oral supplement consisting of 2000 mg daily of C-PAN will be administered to a single cohort of patients.
  Other Names: Calcium Pantothenate; Vitamin B5
Biological: Nivolumab — Nivolumab is an ICI, a type of immunotherapy. It is a monoclonal antibody that binds to the protein PD-1 on the surface of immune cells called T cells. Nivolumab 1 mg/kg every 3 weeks for up to 4 cycles (upon patient´s tolerability) followed by maintenance Nivolumab 3 mg/kg (or fixed dose 240 mg) every 2 weeks or Nivolumab 6 mg/kg (or fixed dose 480 mg) every 4 weeks.
  Other Names: anti-PD-1 antibody
Biological: Ipilimumab — Ipilimumab is an ICI, a type of immunotherapy. It is a monoclonal antibody that binds to the protein CTLA-4 on immune cells called T cells. Ipilimumab 3 mg/kg every 3 weeks for up to 4 cycles.
  Other Names: anti-CLTA-4 antibody

SUMMARY:
This study is open to patients with a type of cancer called melanoma. Patients can join the study if their tumor cannot be removed by surgery or has spread to other organs, and are planned to receive immunotherapy as treatment for their cancer. This study is looking at whether taking calcium pantothenate supplement (a type of Vitamin B5) can increase its levels in the blood and have an effect in the immune system, when its used in combination with the immunotherapy.

DETAILED DESCRIPTION:
This single-center, single-cohort study aims to investigate the effectiveness of oral calcium pantothenate (C-PAN) in raising plasma pantothenic acid levels in melanoma patients. Conducted at Princess Margaret Cancer Centre, the study will enroll 12 eligible subjects with locally unresectable or metastatic melanoma undergoing first-line standard of care (SOC) with combined immune checkpoint inhibitor (ICI) therapy, Nivolumab and Ipilimumab. Additionally, the study will explore changes in immune cell subsets, metabolomics, and gut microbiome to understand the impact of pantothenate/CoA pathway manipulation on ICI efficacy and immune-mediated colitis prevention.

Patients will initially receive a run-in period of C-PAN at a dose of 2000 mg daily for 3 to 7 days, alongside approved SOC drugs. Subsequently, patients will continue with the maintenance dose of 2000 mg daily, starting on the same day as the first cycle of combined ICI. This maintenance dose will be continued until the occurrence of unacceptable toxicity, disease progression by iRECIST criteria, or for a maximum duration of 1 year, whichever comes first, unless there are specific criteria indicating the discontinuation of C-PAN.

For all subjects, radiologic imaging to assess response to treatment will be performed as per standard practice (ideally every 8 to 12 weeks, with first assessment at week 9). Fecal samples will be collected from all subjects at baseline (1st sample), at week 9 following the start of ICI, and at study completion or discontinuation. An additional fecal sample will be collected in case of development of immune-related colitis or immune-related diarrhea.

Standard laboratory investigations for immunotherapy will be collected as per institutional practice. Blood samples for biomarkers will be collected at various time points.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed written and voluntary informed consent.
* 2. Age ≥18 years, male or female.
* 3. Have histologically or cytological documented unresectable stage III or stage IV metastatic melanoma (AJCC 8th edition).
* 4. Have not received any previous systemic treatment for advanced melanoma, including chemotherapy, immunotherapy or targeted therapy.
* 5. Be willing and able to provide stool and blood specimen for analyses at protocol specified time points.
* 6. Performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* 7. Not pregnant for females of child bearing potential as indicated by negative serum or urine pregnancy test within 72 hours of study start

Exclusion Criteria:

* 1. Subjects unable to swallow orally administered medications or any subjects with gastrointestinal disorders likely to interfere with absorption (e.g. bowel obstruction, short gut syndrome, blind loop syndrome, ileostomy, etc.). Subjects with colostomies may be enrolled.
* 2. Subjects with inflammatory bowel disease.
* 3. Any condition that, in the opinion of the Investigator, would interfere with subject safety, or evaluation of the collected specimen and interpretation of study result.
* 4. Pregnant or planning to get pregnant in the next 6 months.
* 5. Female patient breastfeeding.
* 6. Allergy to the investigational product (or its non-medicinal ingredients)- Calcium Pantothenate (stearic acid, Hydroxypropyl methylcellulose) or Immune checkpoint inhibitors (or its non-medicinal ingredients)- Nivolumab (Hydrochloric acid, mannitol (E421), pentetic acid, polysorbate 80, sodium chloride, sodium citrate, sodium hydroxide) and Ipilimumab (diethylene triamine pentaacetic acid (DTPA), mannitol, polysorbate 80, sodium chloride, Tris-hydrochloride, sodium hydroxide, hydrochloric acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To determine if the dose of 2000 mg daily of pantothenic acid achieves an increase in plasmatic concentration of pantothenic acid by at least a 50% between baseline and week 9, in 9 or more of the patients treated with combined ICI. | 9 weeks
  Blood samples will be collected at baseline, and at week 9 to evaluate level in plasmatic pantothenic acid level, measured in mcMol/L.

SECONDARY OUTCOMES:
Evaluate the overall response rate (ORR) of the enrolled cohort. | 1 year
  ORR by RECIST V1.1 and iRECIST.
Evaluate the progression free survival (PFS) of the enrolled cohort. | 1 year
  Measured by RECIST v1.1 and iRECIST.
Incidence of immune-related colitis. | 1 year
  Immune-related colitis will be assessed by CTCAE version 5.
Correlation between baseline intestinal microbiome composition to the development of immune-related colitis. | 1 year
  Correlation between bacteria taxa composition obtained through 16S rRNA sequencing and immune-related colitis.
Correlation between the early changes in composition of intestinal microbiome and the development of immune-related colitis. | 1 year
  Correlate changes in bacteria taxa composition obtained through 16S rRNA sequencing from baseline samples to early time-point (week 9), with the development of immune-related colitis..
The incidence of treatment-related adverse events. | 1 year
  All adverse events that are related to C-PAN and/or in the investigator's opinion is related to immunotherapy will be recorded, and graded as per CTCAE version 5.
The incidence of treatment-related adverse events | 1 year
  Correlation between baseline pantothenic acid plasmatic level in mcMol/L and ORR by RECIST and iRECIST.
Correlation between change in plasmatic pantothenic acid level between baseline and at first day of ICI, and ORR. | 1 year
  Correlation between change in pantothenic acid plasmatic level in mcMol/L between baseline and first day of ICI, and ORR by RECIST and iRECIST.

OTHER OUTCOMES:
Correlation between change in pantothenic acid plasmatic level in mcMol/L between baseline and first day of ICI, and ORR by RECIST and iRECIST. | 2 weeks
  Correlation between change in pantothenic acid plasmatic level in mcMol/L between baseline and first day of ICI, and peripheral blood mononuclear cells examined using flow cytometry, CyTOF and other in vitro immunological assays at first day of ICI.
Correlation between change in plasmatic pantothenic acid level between baseline and week 9 assessment, and immune profiling. | 9 weeks
  Correlation between change in pantothenic acid plasmatic level in mcMol/L between baseline and week 9 assessment, and peripheral blood mononuclear cells examined using flow cytometry, CyTOF and other in vitro immunological assays.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Saibil, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- University Health Network- Princess Margaret Cancer Centre, Toronto, Ontario, Canada